CLINICAL TRIAL: NCT06745739
Title: Life Skills Training Workplace Prevention Program
Acronym: LST-WP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Promotion Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 UDI SP11134-01; 1 UDI SP11134-01 (Other Grant/Funding Number: Substance Abuse and Mental Health Services Administration)
Record Dates: First submitted 2024-12-08; First posted 2024-12-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Job Satisfaction; Work Performance; Health Care Utilization; Depression Symptoms; Stress; Substance Use (Drugs, Alcohol)
MeSH Terms: conditions — Patient Acceptance of Health Care; Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive the Life Skills Training Workplace Prevention Program
  Interventions: Behavioral: Life Skills Training Workplace Prevention Program
- Control (No Intervention): Did not receive the Life Skills Training Workplace Prevention Program

INTERVENTIONS:
Behavioral: Life Skills Training Workplace Prevention Program — A workplace health promotion intervention for youth age 16-24 was adapted from the school-based Life Skills Training program. The program teaches participants the skills necessary to be productive in work and personal settings while also promoting healthy behaviors and preventing or reducing health risk behaviors. Program content focuses on goal-setting and problem-solving skills, stress and anger management skills, effective communication and conflict management skills, time and financial management, substance use risk reduction, and how to contribute to a healthy, safe, and drug-free workplace.
  Arms: Intervention

SUMMARY:
A workplace health promotion intervention for youth age 16-24

DETAILED DESCRIPTION:
A workplace health promotion intervention for youth age 16-24 was adapted from the school-based Life Skills Training program. The program teaches participants the skills necessary to be productive in work and personal settings while also promoting healthy behaviors and preventing or reducing health risk behaviors. Program content focuses on goal-setting and problem-solving skills, stress and anger management skills, effective communication and conflict management skills, time and financial management, substance use risk reduction, and how to contribute to a healthy, safe, and drug-free workplace.

Study Timeline Note: Data collection for this study was conducted between February 2007 and February 2009. The intervention protocols and demographic data reflect the workforce population during this specific timeframe. This registration supports a retrospective analysis of the completed study. While the data are historical, the developmental needs of young adults in the workplace remain relevant.

ELIGIBILITY:
Inclusion Criteria:

* employed at participating store

Exclusion Criteria:

-

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1145 (Actual)
Dates: Start 2007-02-01 (Actual); Primary Completion 2008-08-01 (Actual); Study Completion 2009-02-01 (Actual)

PRIMARY OUTCOMES:
job satisfaction | from baseline assessment up to 18 months post-intervention (assessed at 6-month and 18-month follow-up)
  level of satisfaction with job and frequency of think of about quitting job
work performance | from baseline assessment up to 18 months post-intervention (assessed at 6-month and 18-month follow-up).
  frequency of quality of your work being lower than it should have been, frequency of health problems limiting the kind or amount of work you could do, number of entire workdays missed because of problems with your physical or mental health
health care utilization | from baseline assessment up to 18 months post-intervention (assessed at 6-month and 18-month follow-up).
  saw a medical professional about a work-related injury or illness or about a non-work-related injury or illness
symptoms of depression | from baseline assessment up to 18 months post-intervention (assessed at 6-month and 18-month follow-up).
  frequency of feeling down, depressed, or hopeless; Feeling tired or having little energy; and degree of difficulty for doing your work, take care of things at home, or get along with other people
stress | from baseline assessment up to 18 months post-intervention (assessed at 6-month and 18-month follow-up).
  frequency of being upset because of something that happened unexpectedly; frequency of feeling unable to control the important things in your life; and frequency of finding that you could not cope with all the things you had to do
substance use | from baseline assessment up to 18 months post-intervention (assessed at 6-month and 18-month follow-up)
  frequency of cigarette and tobacco use, alcohol use, illegal drugs

IPD SHARING:
Plan to Share IPD: Yes
The study protocol used in this study is available upon request.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Griffin, K. W., Williams, C., & Botvin, G. J. (2025). Effectiveness of a workplace wellness program for adolescents and young adults. Journal of Workplace Behavioral Health, 1-23.